CLINICAL TRIAL: NCT05048225
Title: Influence of Dietary Salt Intake During Pregnancy on Maternal Systemic and Uteroplacental Vascular Function
Brief Title: Dietary Salt During Pregnancy and Maternal Vascular Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Head of Department of Physiology and Immunology Faculty of Medicine Osijek, Josip Juraj Strossmayer University of Osijek
Other Study IDs: 602-04/21-08/07
Record Dates: First submitted 2021-06-08; First posted 2021-09-17 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Salt; Excess; Pregnancy Related
Keywords: salt intake; microcirculation; macrocirculation; endothelium; uteroplacental function; pregnancy; oxidative stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — serum, placental tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low-salt (LS) group: intake of < 5 g of salt per day
- Normal-salt (NS) group: intake of 5 - 7.5 g of salt per day
- High-salt (HS) group: intake of 7.5 - 10 g of salt per day
- Very high-salt (VHS) group: intake of > 10 g of salt per day

SUMMARY:
The main goal of this study is to investigate the association of dietary salt intake during pregnancy with systemic micro- and macrovascular reactivity and uteroplacental vascular function of the mother, and to examine the potential impact of elevated oxidative stress on this association. Also, the aim is to investigate whether there is an association between excessive salt intake during pregnancy and the outcome of pregnancy.

DETAILED DESCRIPTION:
During the study pregnant women at the third trimester of pregnancy (37-38 weeks of pregnancy) will have one study visit during which following procedures will be done:

* measurement of maternal systemic microvascular function by Laser Doppler flowmetry (post-occlusive reactive hyperemia, iontophoresis of acetylcholine and sodium nitroprusside)
* measurement of maternal systemic macrovascular function by vascular ultrasound measurement of brachial artery flow mediated dilation (FMD)
* measurement of maternal uteroplacental function by ultrasound color Doppler measurement of umbilical artery and fetal middle cerebral artery blood flow
* venous blood sampling; serum will be stored for measurement of oxidative stress, matrix metalloproteinase 9 and endocan level
* 24-hour urine natriuresis (to estimate daily salt intake)
* measurement of blood pressure, heart rate, height and weight, body composition

Immediately after the childbirth following procedures will be done:

* assessment of pregnancy outcome (duration of pregnancy, child birth weight, child birth length and Apgar score)
* placental tissue will be taken and stored for measurement of matrix metalloproteinase 9

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women in the third trimester of pregnancy (37-38 weeks of pregnancy)

Exclusion Criteria:

* smoking
* prenatal hypertension
* thrombophilia
* low molecular weight heparin use
* coronary heart disease
* preconception diabetes
* gestational diabetes
* renal impairment
* cerebrovascular and peripheral artery disease
* any other preconception disease that could affect vascular and endothelial function

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy pregnant women in the third trimester of pregnancy (37-38 weeks of pregnancy)
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal systemic microvascular function | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Skin microvascular reactivity assessed by Laser Doppler flowmetry (post-occlusive reactive hyperemia, iontophoresis of acetylcholine and sodium nitroprusside) - measured in perfusion units (PU)
Maternal systemic macrovascular function | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Vascular ultrasound measurement of brachial artery flow mediated dilation (FMD)
Maternal uteroplacental function | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Ultrasound color Doppler measurement of umbilical artery and fetal middle cerebral artery blood flow

SECONDARY OUTCOMES:
Oxidative stress - thiobarbituric acid reactive substances (TBARS) | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Measurement of biomarkers of oxidative stress level. Thiobarbituric acid reactive substances (TBARS) - biomarker of lipid peroxidation.
Matrix metalloproteinase 9 | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy) (serum) and immediately after childbirth (placental tissue sample)
  ELISA measurement of serum matrix metalloproteinase 9 level in mother serum and placental tissue sample (taken after childbirth)
Endocan | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  ELISA measurement of serum endocan level - proteoglycan associated with endothelium activation
Pregnancy outcome - duration | the outcome measure will be assessed at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Duration of pregnancy (weeks and days)
Pregnancy outcome - birth weight | at one time point immediately after childbirth
  Birth weight (in grams)
Pregnancy outcome - birth length | at one time point immediately after childbirth
  Birth length (in cm)
Pregnancy outcome - Apgar score | at one time point immediately after childbirth
  Apgar score (in Apgar score scale, a total score of 1 to 10; the higher the score, the better the baby is doing after birth)

OTHER OUTCOMES:
Blood pressure | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Automatic oscillometric measurement of systolic and diastolic blood pressure (in mmHg)
Heart rate | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Automatic oscillometric measurement of heart rate (bpm)
Body mass index | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Measurement of BMI (kg/m2)
Body composition | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Body composition and body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Fat Free Mass (FFM kg) and Fat (Fat Mass kg).
Body fluid status | at one time point in the third trimester of pregnancy (37-38 weeks of pregnancy)
  Body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Total Body Water (TBW L), Extracellular Water (ECW L), Intracellular Water (ICW L), Plasma Fluid (PF L) and Interstitial Fluid (IF L).

CONTACTS AND LOCATIONS:
Overall Officials: Ines Drenjancevic, MD, PhD, Study Chair — Faculty of Medicine Josip Juraj Strossmayer University of Osijek
Locations (1):
- Osijek University Hospital, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No